CLINICAL TRIAL: NCT02450669
Title: Practices and Risk Factors for Weaning and Extubation Airway Failure in Adult Intensive Care Unit: a Multicenter Trial
Brief Title: Predictors of Airway Extubation/Weaning Failure
Acronym: Free-Rea
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9242; ID-RCB (Other: 2013-A01402-43)
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Intubation in Intensive Care Units
Keywords: Intubation; Extubation; Weaning; Mechanical ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Airway management in intensive care unit (ICU) patients is challenging. Benefit risk ratio of extubation has to be daily assessed in intubated patients.

The investigators aimed to assess incidence and risk factors of airway failure after extubation procedure in critically ill patients in a prospective multicenter study.

DETAILED DESCRIPTION:
Airway management in intensive care unit (ICU) patients is challenging. Benefit risk ratio of extubation has to be daily assessed in intubated patients. If the patient stay intubated too long, complications of prolonged mechanical ventilation may appear. If the patient is extubated too early, reintubation is associated with higher morbidity and mortality. "Airway failure", defined as the inability to breathe without endotracheal tube, differs from "weaning failure", defined as the inability to breathe spontaneously without invasive mechanical ventilation. "Mixed failure" occurs when extubation failure is caused by both airway and weaning failure. However, most of the studies assessing criteria of success of extubation did not separate airway from weaning success.

Study design and population A prospective, observational, multicenter study will be conducted in ICUs to develop a predictive model for airway failure following extubation. All adult patients consecutively intubated in ICU will be included. Exclusion criteria are pregnancy, refusal to participate after information was provided or age under 18 years old.

Ethics and consent Because of the observational, non invasive design of this study, the need for written consent is waived. The local ethics committee "Comité de Protection des personnes Sud-Mediterranée III" approved the study design (code UF: 9242, register: 2013-A01402-43).

Data collection Clinical parameters will be prospectively assessed before, during and after extubation procedure. In summary, the following data will be assessed before extubation : demographic data, body mass index (BMI), severity scores (Simplified Acute Physiologic Score (SAPS) II at admission, Sequential Organ Failure Assessment (SOFA) score on the day of the procedure), type of admission (medical vs surgical), co morbidities such as ethylism, smoking, cirrhosis, chronic obstructive pulmonary disease (COPD), cause of admission, cause and location of initial intubation, hypotension episode during the stay, difficulty of intubation, material used for intubation, Mallampati score, Cormack score, date and hour of extubation, a previous intubation in the last two weeks. Will be also assessed before extubation the type of spontaneous breathing trial (SBT), the use of a weaning mode before extubation, standard analysis, physiotherapy measurements, the assessment of agitation and answer to simple orders, the strength of cough, the perception of the extubation by the patient, a leak test before extubation, the blood results at the end of the SBTs, the succion rate and secretions aspect, the use of systemic corticotherapy before extubation.

Just before and during the extubation, sequential organ failure assessment (SOFA) score will be assessed, as the information of the patient, the nature and number of the operators, preoxygenation before extubation, precautions used in case of extubation failure.

Just after extubation, will be assessed physiotherapy after extubation, aerosols of corticoids or adrenalins post extubation, and the occurrence in the hour after extubation of complications. At 48 hours post extubation, the occurrence of reintubation will be evaluated, and its relation with airway failure, weaning failure, or both (mixed failure). In case of reintubation, the delay between extubation and reintubation will be informed, and the cause of reintubation. Finally, at ICU discharge, the mortality will be analyzed, the occurrence of late reintubation (>48h), the use and the length of mechanical or non invasive ventilation, the need for vasopressors or dialysis after extubation, the occurrence of a nosocomial pneumonia, a catheter infection, a bacteremia, a urinary infection. At the exit of the hospital, the mortality at day 28 following extubation will be assessed.

Definition of extubation failure, airway failure, weaning failure, mixed failure and complications Extubation failure is defined as the need to reintubate less than 48 hours after extubation. The need to reintubate was left to the physician appreciation in this observational study. Airway failure is defined as an extubation failure because of the inability to breathe without a tracheal tube. Weaning failure is defined as an extubation failure because of the inability to breathe without an invasive mechanical ventilation. Mixed failure is a combination of airway and weaning failure. Severe life-threatening complications are defined as death, cardiac arrest, severe cardiovascular collapse, defined as systolic blood pressure<65 mmHg recorded at least one time and/or <90 mmHg that lasted 30min despite 500-1,000 ml of fluid loading (crystalloids/or colloids solutions) and/or requiring introduction of vasoactive support, or severe hypoxemia (decrease in SpO2 below 80% during attempts), occurring during the first hour following intubation.

Outcomes The primary outcome are the risk factors for airway failure following extubation. The secondary outcomes are the risk factors of extubation failure, weaning failure and mixed failure, the incidence of extubation failure, airway failure, weaning failure and mixed failure, the severe life-threatening complications related to extubation in ICU, the moderate complications related to extubation in ICU, the rate of difficult intubation in case of extubation failure.

Statistical analysis Quantitative variables will be expressed as means (standard deviation) or medians (interquartiles 25%-75%) and compared using the student t test or the Wilcoxon test as appropriate (Gaussian or non Gaussian variables). Qualitative variables will be compared using the chi 2 test or the Fisher test as appropriate.

A logistic regression will be used to identify risk factors of airway failure. A multivariate model will be established.

A p-value of < and = 0.05 will be considered statistically significant. The statistical analysis will be performed by the medical statistical department of the Montpellier University Hospital with the help of statistical software (SAS, version 9.3; SAS Institute; Cary, NC and R, version 2.14.1).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient extubated in the ICU

Exclusion Criteria:

* Decision not to reintubate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the adult patients extubated in the ICU
Sampling Method: Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2013-12-19 (Actual); Primary Completion 2015-07-04 (Actual); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
Risk factors of airway failure (logistic regression will be used to identify risk factors) | 48 hours

SECONDARY OUTCOMES:
Risf factors of extubation failure and weaning failure (Quantitative variables will be expressed as means (standard deviation) or medians (interquartiles 25%-75%) and compared using the student t test or the Wilcoxon test as appropriate | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Samir JABER, PU-PH, Principal Investigator — Hospital of Montpellier
Locations (1):
- CHU Montpellier, Montpellier, France

REFERENCES:
- [Result] Marini JJ, Smith TC, Lamb VJ. External work output and force generation during synchronized intermittent mechanical ventilation. Effect of machine assistance on breathing effort. Am Rev Respir Dis. 1988 Nov;138(5):1169-79. doi: 10.1164/ajrccm/138.5.1169. PMID 3202477
- [Result] Moschietto S, Doyen D, Grech L, Dellamonica J, Hyvernat H, Bernardin G. Transthoracic Echocardiography with Doppler Tissue Imaging predicts weaning failure from mechanical ventilation: evolution of the left ventricle relaxation rate during a spontaneous breathing trial is the key factor in weaning outcome. Crit Care. 2012 May 14;16(3):R81. doi: 10.1186/cc11339. PMID 22583512
- [Result] Montgomery AB, Holle RH, Neagley SR, Pierson DJ, Schoene RB. Prediction of successful ventilator weaning using airway occlusion pressure and hypercapnic challenge. Chest. 1987 Apr;91(4):496-9. doi: 10.1378/chest.91.4.496. PMID 3829740
- [Result] Epstein SK, Ciubotaru RL. Independent effects of etiology of failure and time to reintubation on outcome for patients failing extubation. Am J Respir Crit Care Med. 1998 Aug;158(2):489-93. doi: 10.1164/ajrccm.158.2.9711045. PMID 9700126
- [Result] Witt NJ, Zochodne DW, Bolton CF, Grand'Maison F, Wells G, Young GB, Sibbald WJ. Peripheral nerve function in sepsis and multiple organ failure. Chest. 1991 Jan;99(1):176-84. doi: 10.1378/chest.99.1.176. PMID 1845860
- [Result] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Result] Annane D, Sebille V, Charpentier C, Bollaert PE, Francois B, Korach JM, Capellier G, Cohen Y, Azoulay E, Troche G, Chaumet-Riffaud P, Bellissant E. Effect of treatment with low doses of hydrocortisone and fludrocortisone on mortality in patients with septic shock. JAMA. 2002 Aug 21;288(7):862-71. doi: 10.1001/jama.288.7.862. PMID 12186604
- [Result] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Result] Epstein SK, Ciubotaru RL, Wong JB. Effect of failed extubation on the outcome of mechanical ventilation. Chest. 1997 Jul;112(1):186-92. doi: 10.1378/chest.112.1.186. PMID 9228375
- [Result] Rothaar RC, Epstein SK. Extubation failure: magnitude of the problem, impact on outcomes, and prevention. Curr Opin Crit Care. 2003 Feb;9(1):59-66. doi: 10.1097/00075198-200302000-00011. PMID 12548031
- [Result] Francon D, Jaber S, Pean D, Bally B, Marciniak B. [Difficult extubation: extubation criteria and management of risk situations: question 6. Societe Francaise d'Anesthesie et de Reanimation]. Ann Fr Anesth Reanim. 2008 Jan;27(1):46-53. doi: 10.1016/j.annfar.2007.10.026. Epub 2007 Dec 31. No abstract available. French. PMID 18164897
- [Result] Jaber S, Chanques G, Matecki S, Ramonatxo M, Vergne C, Souche B, Perrigault PF, Eledjam JJ. Post-extubation stridor in intensive care unit patients. Risk factors evaluation and importance of the cuff-leak test. Intensive Care Med. 2003 Jan;29(1):69-74. doi: 10.1007/s00134-002-1563-4. Epub 2002 Nov 22. PMID 12528025
- [Result] Tanaka A, Isono S, Ishikawa T, Nishino T. Laryngeal reflex before and after placement of airway interventions: endotracheal tube and laryngeal mask airway. Anesthesiology. 2005 Jan;102(1):20-5. doi: 10.1097/00000542-200501000-00007. PMID 15618782
- [Result] Jaber S, Jung B, Matecki S, Petrof BJ. Clinical review: ventilator-induced diaphragmatic dysfunction--human studies confirm animal model findings! Crit Care. 2011 Mar 11;15(2):206. doi: 10.1186/cc10023. PMID 21457528
- [Result] Jaber S, Petrof BJ, Jung B, Chanques G, Berthet JP, Rabuel C, Bouyabrine H, Courouble P, Koechlin-Ramonatxo C, Sebbane M, Similowski T, Scheuermann V, Mebazaa A, Capdevila X, Mornet D, Mercier J, Lacampagne A, Philips A, Matecki S. Rapidly progressive diaphragmatic weakness and injury during mechanical ventilation in humans. Am J Respir Crit Care Med. 2011 Feb 1;183(3):364-71. doi: 10.1164/rccm.201004-0670OC. Epub 2010 Sep 2. PMID 20813887
- [Derived] Aarab Y, Pensier J, Garnier F, Monet C, Lakbar I, Chanques G, de Jong A, Capdevila M, Jaber S; FreeRea study group. Incidence and outcomes of extubation failure in mechanically ventilated patients with cirrhosis: a post-hoc analysis of a prospective multicenter study. Ann Intensive Care. 2025 Oct 16;15(1):160. doi: 10.1186/s13613-025-01576-3. PMID 41099917
- [Derived] De Jong A, Capdevila M, Aarab Y, Cros M, Pensier J, Lakbar I, Monet C, Quintard H, Cinotti R, Asehnoune K, Arnal JM, Guitton C, Paugam-Burtz C, Abback P, Mekontso-Dessap A, Lakhal K, Lasocki S, Plantefeve G, Claud B, Pottecher J, Corne P, Ichai C, Molinari N, Chanques G, Papazian L, Azoulay E, Jaber S; FREE-REA Study Group. Incidence, Risk Factors, and Long-Term Outcomes for Extubation Failure in ICU in Patients With Obesity: A Retrospective Analysis of a Multicenter Prospective Observational Study. Chest. 2025 Jan;167(1):139-151. doi: 10.1016/j.chest.2024.07.171. Epub 2024 Sep 7. PMID 39182573
- [Derived] Jaber S, Quintard H, Cinotti R, Asehnoune K, Arnal JM, Guitton C, Paugam-Burtz C, Abback P, Mekontso Dessap A, Lakhal K, Lasocki S, Plantefeve G, Claud B, Pottecher J, Corne P, Ichai C, Hajjej Z, Molinari N, Chanques G, Papazian L, Azoulay E, De Jong A. Risk factors and outcomes for airway failure versus non-airway failure in the intensive care unit: a multicenter observational study of 1514 extubation procedures. Crit Care. 2018 Sep 23;22(1):236. doi: 10.1186/s13054-018-2150-6. PMID 30243304